CLINICAL TRIAL: NCT05167318
Title: Frequent Standardized Oral Care to Improve Health Outcomes in Premature Infants in the Neonatal Intensive Care Unit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202101340
Record Dates: First submitted 2021-11-18; First posted 2021-12-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Microbial Colonization; Ventilator Associated Pneumonia
MeSH Terms: conditions — Communicable Diseases; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- every 3-4 hour oral care (Experimental): Infants will receive standardized oral care every 3-4 hours for 4 weeks
  Interventions: Other: frequent standardized oral care
- every 12 hour oral care (No Intervention): Infants will receive standardized oral care every 12 hours for 4 weeks

INTERVENTIONS:
Other: frequent standardized oral care — Standardized oral care will be provided every 3-4 hours
  Arms: every 3-4 hour oral care

SUMMARY:
Premature very low birth weight (VLBW) infants are susceptible to complications related to infrequent and non-standardized oral care. Although the benefits of frequent standardized oral care are known to reduce oral dybiosis (increased level of potentially pathogenic bacteria) and its associated complications in critically ill adults leading to established evidence-based guidelines, no such information exists for VLBW infants. The proposed study will prospectively follow 40 VLBW infants for 4 weeks following birth. Infants will be randomized into 1 of 2 groups. Standardized oral care will be performed every 3-4 hours (Group 1) and every 12 hours (Group 2). Aim 1 will evaluate the feasibility of frequent standardized oral care, Aim 2 will compare the oral microbiome between groups, and Aim 3 will compare respiratory outcomes including the incidence of ventilator associated pneumonia, bronchopulmonary dysplasia and need for respiratory support between infants receiving standardized oral care every 3-4 hours and every 12 hours. Issues related to recruitment, retention, randomization, acceptance by nursing staff, and treatment fidelity will be examined. Saliva samples will be obtained weekly and analyzed using 16S sequencing, respiratory cultures will be obtained weekly on ventilated infants, and respiratory outcomes will be collected from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 weeks
* birth weight < 1500 grams
* mother is English speaking
* mother is > 18 years of age.

Exclusion Criteria:

* Congenital anomalies of the face, lungs, or gastrointestinal system
* not expected to survive

Ages: 12 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Type of of bacterial in the oral cavity | weekly for 4 weeks
  microbial analysis of the oral microbiome

SECONDARY OUTCOMES:
Days of respiratory support | Up to 100 days
  number of days infant was on respiratory support
Incidence of chronic lung disease | Up to 100 days
  Whether or not the infant was diagnosed with chronic lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Parker, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No